CLINICAL TRIAL: NCT03431688
Title: Efficacy Comparison of Metronidazole-based Triple and Bismuth-based Quadruple Therapy for Clarithromycin Resistant-Helicobacter Pylori Infection: Randomized Controlled Trial
Brief Title: Tailored Therapy for Clarithromycin-Resistant H. Pylori
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangdong Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Shin, Woon Geon, Woon Geon Shin, Kangdong Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KangdongSHH
Record Dates: First submitted 2018-01-31; First posted 2018-02-13 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2022-04

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PAM (Active Comparator): treatment with PPI, metonidazole, amoxicillin
  Interventions: Drug: PAM
- PBMT (Active Comparator): treatment with PPI, metonidazole, bismuth, tetracyclin
  Interventions: Drug: PBMT

INTERVENTIONS:
Drug: PAM — treatment with PPI, metonidazole, amoxicillin
  Arms: PAM
Drug: PBMT — treatment with PPI, metonidazole, bismuth, tetracyclin
  Arms: PBMT

SUMMARY:
Clarithromycin-resistant H. pylori is the main cause of H. pylori eradication failure. Tailored therapy on the basis of detection of a clarithromycin resistance mutation by PCR has been studied recently, however, there have been few studies comparing treatment regimen in patient with clarithromycin-resistant H. pylori. We used sequencing-based clarithromycin resistance mutation and aimed to compare PAM (proton pump inhibitor, amoxicilline, metronidazole) regimen and PBMT (proton pump inhibitor, bismuth, metronidazole, tetracyclin) regimen in patient with clarithromycin-resistant H. pylori.

ELIGIBILITY:
Inclusion Criteria:

* peptic ulcer disease
* H. pylori gastritis
* low grade MALT lymphoma

Exclusion Criteria:

* history of gastric cancer surgery
* severe comorbidity (ESRD, LC)
* hypersensitivity to drug
* pregnancy

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 782 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
H. pylori eradication rate | 14 days
  H. pylori eradication rate

CONTACTS AND LOCATIONS:
Overall Officials: Woon Geon Shin, Principal Investigator — Kangdong Sacred Heart Hospital
Locations (1):
- Kangdong Sacred Heart Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No